CLINICAL TRIAL: NCT03791034
Title: Prospective Feasibility Study of Cell Free Circulating Tumor DNA for the Diagnosis and Treatment Monitoring in Early-stage Non-small Cell Lung Cancer
Brief Title: Cell Free DNA for the Diagnosis and Treatment in Early NSCLC
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Guardant Health, Inc. (Industry)
Responsible Party: Principal Investigator, Jhingook Kim, MD, Professor, Samsung Medical Center
Other Study IDs: 2017-08-041-003
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Recurrence; cfDNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect peripheral blood cell-free tumor DNA serially in non-small cell lung cancer cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate whether peripheral circulating cell-free tumor DNA (cfDNA) can aid screening of recurrence after complete resection of early stage non-small cell lung cancer.

DETAILED DESCRIPTION:
During evolution of primary tumor, tumor cells can be released into the bloodstream. It has also been shown that circulating cell-free tumor DNA (cfDNA) is released from apoptotic or necrotic tumor cells. In a study of cfDNA level after surgery in colon cancer patients, they suggested that cfDNA could detect recurrence of cancer several months earlier than the conventional follow up studies. Following several reports have suggested that cfDNA can invade host cells and alter host cell biology to cause cancer metastasis.

In this regard, we will collect from non-small cell lung cancer patients cohort who underwent curative resection, and will evaluate whether peripheral cfDNA can aid early detection of cancer recurrence. We will also study the genomic signature of cfDNA to assess the relationship between cfDNA and clinical outcome of non-small cell lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* All subjects need to sign the informed consent form
* All subjects have Non-small cell lung cancer which suspected on chest CT or confirmed pathologically preoperatively.
* Non-small cell lung cancer have to confirmed pathologically after operation
* Clinical stage I - IIIA by AJCC 7th staging system

Exclusion Criteria:

* Have been undergone chemotherapy or radiotherapy due to non-small call lung cancer
* Have been diagnosed any type of cancer other than cancer of skin, thyroid, uterine cervix with 3 years before enrollment
* Recurrent lung cancer
* Stage IIIB, IV by AJCC 7th staging system

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-small cell lung cancer patients who undergone curative surgery
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 24 months
  Recurrence of primary tumor documented by diagnostic imaging with or without biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jhingook Kim, MD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No